CLINICAL TRIAL: NCT00877032
Title: A Phase I, Double-masked, Placebo-controlled Study Evaluating The Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, And Immunogenicity Of Single Escalating Doses Of Rn6g In Patients With Dry, Age-related Macular Degeneration (Amd)
Brief Title: Safety And Tolerability Study Of RN6G In Patients With Dry, Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1181001
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Age-Related Maculopathy; Age-Related Maculopathies; Eye Diseases; Retinal Degeneration; Macular Degeneration
Keywords: Phase 1; Dry Age Related Macular Degeneration; RN6G
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Retinal Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: RN6G; Biological: Placebo

INTERVENTIONS:
Biological: RN6G — intravenous, single dose, dose ranging from 0.3mg/kg up to a maximum of 40 mg/kg.
Biological: Placebo — intravenous, single dose with experimental dose.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of RN6G in patients with dry, age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Be of non-childbearing potential.
* Diagnosis of dry AMD as defined by the Age-Related Eye Disease Study (AREDS, 2005), including uni- or multi-focal GA, without foveal involvement.
* BCVA of 20/320 or better in the worst eye.

Exclusion Criteria:

* Diagnosis of exudative (wet) AMD, with subretinal or choroidal neovascular lesions.
* Diagnosis or history of Alzheimer's disease, dementia or neurodegenerative disorders.
* Diagnosis or recent history of clinically significant cerebrovascular disease.
* Uncontrolled hypertension.
* Uncontrolled Type 1 or Type 2 diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Dedicated Phase 1, Phoenix, Arizona
  - Retinal Consultants of AZ, Phoenix, Arizona
  - Insight Diagnostic Imaging Center, Phoenix, Arizona
  - Amir Hedayati-Rad, MD, Glendale, California
  - United Medical Imaging, Inglewood, California
  - United Medical Research Institute, Inglewood, California
  - California Pharmacy and Compounding Center, Newport Beach, California
  - Jasper Clinic, Inc., Kalamazoo, Michigan
  - Jonathan Rowe, MD, Kalamazoo, Michigan
  - Ronald VanderLugt, MD, Kalamazoo, Michigan
  - CEDRA Clinical Research, LLC, San Antonio, Texas
  - Village Drive Imaging Center, San Antonio, Texas
  - Specialty MRI, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - EZ Pass Rx, Bountiful, Utah
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Rocky Mountain Eye Care Associates, LC, Salt Lake City, Utah
  - Western Neurological Associates, Salt Lake City, Utah

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1181001&StudyName=Safety%20And%20Tolerability%20Study%20Of%20RN6G%20In%20Patients%20With%20Dry%2C%20Age-Related%20Macular%20Degeneration

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From a given cohort, no more than 3 participants received treatment on Day 1, the remaining participants in the respective cohort received treatment at least 24 hours thereafter. All the remaining participants were treated on same day, if required, as per site scheduling.
Groups:
- RN6G 0.3 mg/kg: Single intravenous infusion dose of RN6G 0.3 milligram per kilogram (mg/kg) of body weight over 120 to 160 minutes on Day 1.
- RN6G 1 mg/kg: Single intravenous infusion dose of RN6G 1 mg/kg of body weight over 120 to 160 minutes on Day 1.
- RN6G 3 mg/kg: Single intravenous infusion dose of RN6G 3 mg/kg of body weight over 120 to 160 minutes on Day 1.
- RN6G 10 mg/kg: Single intravenous infusion dose of RN6G 10 mg/kg of body weight over 120 to 160 minutes on Day 1.
- RN6G 20 mg/kg: Single intravenous infusion dose of RN6G 20 mg/kg of body weight over 120 to 160 minutes on Day 1.
- RN6G 40 mg/kg: Single intravenous infusion dose of RN6G 40 mg/kg of body weight over 120 to 160 minutes on Day 1.
- Placebo: Single intravenous infusion dose of placebo matched to RN6G on Day 1.
Period: Overall Study
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo
Started | 6 | 6 | 6 | 7 | 6 | 6 | 20
Treated | 6 | 6 | 6 | 6 | 6 | 6 | 18
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 18
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Did not meet entrance criteria | 0 | 0 | 0 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received any amount of the single dose of either study drug or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (11.1) | 70.2 (9.9) | 65.5 (10.4) | 69.2 (3.7) | 67.8 (7.5) | 65.0 (6.5) | 67.4 (8.2) | 67.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 2 | 5 | 4 | 14 | 36
  Male | 2 | 4 | 1 | 4 | 1 | 2 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular Adverse Events (AEs)
Description: AE: untoward medical occurrence in participant who received study drug without regard to causal relationship. Ocular AE was identified by spontaneous report or ocular examination: early treatment diabetic retinopathy study (ETDRS) best-corrected visual acuity (BCVA); low-luminance BCVA; pupillary light response, extra-ocular muscle movements, external examination of the eyelids and eyelashes, slit-lamp biomicroscopic examination (SLE) of all components of the anterior and posterior segments, intra-ocular pressure (IOP), and dilated ocular fundus examination of the vitreous and retina. AE was assessed according to severity; mild (did not interfere with participant's usual function), moderate (interfered to some extent with participant's usual function) and severe (interfered significantly with participant's usual function). Total number of participants with ocular (related to eye) AEs and severity was reported.
Time Frame: Baseline up to Day 168
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 18
participants
  Ocular AEs | 1 | 3 | 2 | 1 | 4 | 3 | 6
  Mild ocular AEs: right eye | 1 | 1 | 1 | 0 | 1 | 0 | 2
  Mild ocular AEs: left eye | 1 | 2 | 1 | 0 | 1 | 2 | 2
  Mild ocular AEs: both eyes | 0 | 1 | 1 | 1 | 2 | 1 | 3
  Moderate ocular AEs: right eye | 1 | 1 | 1 | 0 | 1 | 0 | 1
  Moderate ocular AEs: left eye | 1 | 0 | 0 | 0 | 2 | 0 | 1
  Moderate ocular AEs: both eyes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe ocular AEs: right eye | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe ocular AEs: left eye | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe ocular AEs: both eyes | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Incidence and Severity of Systemic Adverse Events (AEs)
Description: AE: untoward medical occurrence in participant who received study drug without regard to causal relationship. Systemic AEs was identified by spontaneous report or physical and neurological examinations changes in vital signs, clinical laboratory abnormalities, 12-lead electrocardiograms (ECG), brain magnetic resonance imaging (MRI). AE was assessed according to severity; mild (did not interfere with participant's usual function), moderate (interfered to some extent with participant's usual function) and severe (interfered significantly with participant's usual function). Total number of participants with systemic (all AEs including eye-related) AEs and severity was reported.
Time Frame: Baseline up to Day 168
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 18
participants
  Systemic AEs | 4 | 5 | 5 | 4 | 6 | 6 | 15
  Mild systemic AEs | 4 | 5 | 5 | 2 | 6 | 5 | 15
  Moderate systemic AEs | 1 | 2 | 2 | 2 | 3 | 2 | 7
  Severe systemic AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - Inf)] of RN6G
Description: AUC (0 - inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf). Participants who received RN6G were reported.
Time Frame: Pre-dose on Day 1; 1 hour (hr) during infusion on Day 1; 0, 1, 4, 8, 12 hrs post-dose on Day 1; Day 2, 7, 14, 21, 28, 42, 56, 84, 168
Population: Pharmacokinetic (PK) analysis population included all participants who received any amount of the single dose of RN6G. Here "N" (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: microgram*hour/milliliter (mcg*hr/mL)
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
microgram*hour/milliliter (mcg*hr/mL) | 1003 (399) | 4516 (627) | 19591 (3657) | 76987 (18255) | 163049 (57995) | 486191 (64822)

4. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of RN6G
Description: AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t). Participants who received RN6G were reported.
Time Frame: as for outcome 3
Population: PK analysis population included all participants who received any amount of the single dose of RN6G.
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
mcg*hr/mL | 836 (326) | 3990 (593) | 17878 (3395) | 72792 (15929) | 155377 (52319) | 472239 (59181)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of RN6G
Description: Participants who received RN6G were reported.
Time Frame: as for outcome 3
Population: PK analysis population included all participants who received any amount of the single dose of RN6G.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
mcg/mL | 4.70 (0.87) | 23.1 (2.9) | 75.2 (9.3) | 286 (58) | 435 (87) | 1245 (142)

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of RN6G
Description: Participants who received RN6G were reported.
Time Frame: as for outcome 3
Population: PK analysis population included all participants who received any amount of the single dose of RN6G.
Measure: Median (Full Range); unit: hours
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hours | 2.1 [2.0 to 3.3] | 2.1 [2.0 to 3.1] | 2.0 [2.0 to 6.2] | 4.5 [3.0 to 14.2] | 2.5 [2.1 to 10.0] | 2.1 [2.0 to 6.0]

7. Secondary Outcome: Volume of Distribution (Vd) of RN6G
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Participants who received RN6G were reported and volume was measured as volume/kg of body weight.
Time Frame: as for outcome 3
Population: PK analysis population included all participants who received any amount of the single dose of RN6G. Here "N" (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mL/kilogram (mL/kg)
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
mL/kilogram (mL/kg) | 384 (86.8) | 555 (180) | 336 (74.8) | 230 (39.5) | 198 (57.1) | 98.0 (12.1)

8. Secondary Outcome: Clearance (CL) of RN6G
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. Participants who received RN6G were reported and clearance was measured as mL/hr/kg of body weight.
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
mL/hr/kg | 0.336 (0.117) | 0.225 (0.0287) | 0.158 (0.031) | 0.137 (0.037) | 0.134 (0.040) | 0.0835 (0.0115)

9. Secondary Outcome: Mean Residence Time (MRT) of RN6G
Description: MRT was calculated as area under the moment curve from time 0 to extrapolated infinite time (AUMC[0 to inf])/area under the concentration effect curve from time 0 to extrapolated infinite time (AUC[0 to inf]). AUMC (0 to inf)= area under the moment curve from 0 to time t (AUMC 0-t) + [(Ct*tlast )/lamdaz ] + [Ct/(lamdaz )^2 ] where Ct= last measurable concentration, tlast= last measurable time, lamdaz= apparent terminal elimination rate constant. Participants who received RN6G were reported.
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
days | 36.2 (19.7) | 57.3 (16.8) | 51.5 (5.8) | 37.7 (8.3) | 41.9 (10.0) | 38.0 (6.8)

10. Secondary Outcome: Plasma Terminal Half-life (t1/2) of RN6G
Description: Plasma terminal half-life is the time measured for the plasma concentration to decrease by one half. Participants who received RN6G were reported.
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
days | 37.5 (20.1) | 71.5 (20.5) | 61.4 (5.8) | 50.1 (9.4) | 43.3 (6.7) | 34.2 (5.1)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Amyloid (A) Beta(1-X)
Time Frame: as for outcome 3
Population: Pharmacodynamic (PD) analysis population included all participants who received any amount of the single dose of either study drug or placebo.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 18
picogram/milliliter (pg/mL) | 3607 (1517) | 10318 (3312) | 21267 (2836) | 59000 (14599) | 70967 (10265) | 75700 (11773) | 533 (177)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Amyloid (A) Beta(1-X)
Time Frame: as for outcome 3
Population: PD analysis population included all participants who received any amount of the single dose of either study drug or placebo.
Measure: Median (Full Range); unit: hours
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 18
hours | 14.3 [6.3 to 27.0] | 26.0 [14.1 to 26.0] | 26.1 [23.9 to 149] | 160 [148 to 461] | 317 [169 to 651] | 402 [270 to 1330] | 14.3 [1.0 to 4012]

13. Secondary Outcome: Area Under the Curve From Time Zero to Day 165 [AUC (0-165d)] of Amyloid (A) Beta(1-X)
Description: AUC (0-165d)= Area under the plasma concentration versus time curve from time zero (pre-dose) to Day 165.
Time Frame: Pre-dose on Day 1; 1 hour (hr) during infusion on Day 1; 0, 1, 4, 8, 12 hrs post-dose on Day 1; Day 2, 7, 14, 21, 28, 42, 56, 84, 165
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram*hr/mL (ng*hr/mL)
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 18
nanogram*hr/mL (ng*hr/mL) | 2512 (752) | 4512 (1780) | 12041 (2553) | 46852 (12562) | 85441 (22829) | 113547 (19280) | 1572 (392)

14. Secondary Outcome: Number of Participants With Anti-Drug Anti-body
Description: Participants tested positive for anti-drug anti-body on at least one or more occasions were reported.
Time Frame: Baseline up to Day 168
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 18
participants | 2 | 1 | 0 | 2 | 1 | 2 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | RN6G 0.3 mg/kg | RN6G 1 mg/kg | RN6G 3 mg/kg | RN6G 10 mg/kg | RN6G 20 mg/kg | RN6G 40 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/18
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 5/6 | 4/6 | 6/6 | 6/6 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RN6G 0.3 mg/kg (N=6) | RN6G 1 mg/kg (N=6) | RN6G 3 mg/kg (N=6) | RN6G 10 mg/kg (N=6) | RN6G 20 mg/kg (N=6) | RN6G 40 mg/kg (N=6) | Placebo (N=18)
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RN6G 0.3 mg/kg (N=6) | RN6G 1 mg/kg (N=6) | RN6G 3 mg/kg (N=6) | RN6G 10 mg/kg (N=6) | RN6G 20 mg/kg (N=6) | RN6G 40 mg/kg (N=6) | Placebo (N=18)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract cortical (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 3
Cataract nuclear (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iritis (Eye disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pupillary disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal pigment epitheliopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity tests abnormal (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 1 | 4 | 2 | 3
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Results for pharmacodynamic parameters [Cmax, Tmax and AUC (0-65d) of A beta(1-X)], are presented as absolute values at specified time points and not as change from baseline as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.